CLINICAL TRIAL: NCT02034149
Title: The Cost Effectiveness and Evaluation of Disease Management of Chronic Kidney Disease and High Risk Population
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Collaborators: Ministry of Health and Welfare, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DMR100-IRB-206
Record Dates: First submitted 2013-11-29; First posted 2014-01-13 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-07

CONDITIONS: Chronic Kidney Diseases; Chronic Kidney Insufficiency
Keywords: chronic kidney disease; high risk; intervention; hypertension; hyperglycemia; hyperlipidemia
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension; Hyperglycemia; Hyperlipidemias | interventions — Self-Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- general management (Other): All participants received a general education with the knowledge on care for early chronic kidney disease recently establishes by the National Health Insurance system. We then used the cross-theoretical model to assess the intervention among the three groups.We collected information on baseline and follow-up data on biochemical and physiological check-ups, health promotion behavior, dietary intake status, self-efficacy and cost etc. The effectiveness assessments have been set for the baseline, 3rd, 6th, 12th and 18th months.
  Interventions: Behavioral: general management
- self-management (Experimental): Participants in the self-management group are expected to emphasize on self-managed interventions, including self-monitoring and records keeping, self-education with digital video disc (DVD) courses. We negotiated their behavior change set goals for them etc.With one year of intervention period, the 3 groups will be assessed at the 18th months of follow-up next year.
  Interventions: Behavioral: general management; Behavioral: self-management
- peer-assisted management (Experimental): The peer-assisted management group received the peer oriented group activities followed, including group discussions to share experience and sports map etc. With one year of intervention period, the 3 groups will be assessed at the 18th months of follow-up next year.
  Interventions: Behavioral: general management; Behavioral: self-management; Behavioral: peer-assisted management

INTERVENTIONS:
Behavioral: general management — All participants received a general education with the knowledge on care for early chronic kidney disease recently establishes by the National Health Insurance system. We then used the cross-theoretical model to assess the intervention among the three groups.
  Other Names: A general education.
Behavioral: self-management — Participants in the self-management group are expected to emphasize on self-managed interventions, including self-monitoring and records keeping, self-education with DVD courses. We negotiated their behavior change set goals for them etc.
  Other Names: Self-managed interventions.
  Arms: peer-assisted management; self-management
Behavioral: peer-assisted management — The peer-assisted management group received similar program for 3 months, the peer oriented group activities followed, including group discussions to share experience and sports map etc.
  Other Names: the peer oriented group activities.
  Arms: peer-assisted management

SUMMARY:
This study is being implemented for 3 aims. The first has been to conduct a systematic literatures review on CKD intervention models and their effectiveness. Findings have been adopted in our intervention program. The second purpose is to establish a practical management model or an intervention model for CKD patients and high risk population with the 18-month of follow-up.In the third year, we will use social perspective point to evaluate the costs and the benefits of intervention.

DETAILED DESCRIPTION:
The object of the study is by screening for adults (20 years) with chronic kidney disease (CKD stage 1-3a) and high-risk groups. They were randomly assigned into experimental groups (self management and peer-assisted management) and control group (general management). All participants received a general education with the knowledge on care for early chronic kidney disease recently establishes by the National Health Insurance system. We then used the cross-theoretical model to assess the intervention among the three groups.

We collected information on baseline and follow-up data on biochemical and physiological check-ups, health promotion behavior, dietary intake status, self-efficacy and cost etc. Information on behavior changes, including smoking, chewing betel nut, medication, exercise and diet, was also collected and assessed. Participants in the self-management group are expected to emphasize on self-managed interventions, including self-monitoring and records keeping, self-education with digital video disc (DVD) courses. We negotiated their behavior change set goals for them etc. The peer-assisted management group received similar program for 3 months, the peer oriented group activities followed, including group discussions to share experience and sports map etc. The effectiveness assessments have been set for the baseline, 3rd, 6th, 12th and 18th months. With one year of intervention period, the 3 groups will be assessed at the 18th months of follow-up next year.

In the third year, we will use social perspective point to evaluate the costs and benefits of intervention. We suppose that a 100,000 people to screen out cases of chronic kidney disease (CKD stage 1-3a) and high-risk groups, and we will compare the cost-effectiveness analysis between the experimental group with accept the intervention for 12 months to the control groups without receiving extra intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 20 with chronic kidney disease (CKD) stage 1-3a patients and high-risk groups.

Exclusion Criteria:

* Inability to communicate in Chinese.
* Lack of capacity to write in Chinese.
* Ongoing treatment in dialysis.
* Suffering from major diseases.
* Treatment in cancer or suffering from cancer less than two years.
* Have received organ transplants or bone marrow transplantation.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 411 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Renal function at 18 months | the baseline, 3rd, 6th, 12th and 18th months.

SECONDARY OUTCOMES:
Achievement of self management in drug compliance,exercise habit,balance diet at 18 months | the baseline, 3rd, 6th, 12th and 18th months.

OTHER OUTCOMES:
Compliance to educational programs(exercise, drug, diet) in 18 months | 18th months.

CONTACTS AND LOCATIONS:
Overall Officials: Chiu-Ching Huang, doctor, Study Director — Department of Medicine
Locations (1):
- China Medical University Hospital, Taichung, Taiwan